CLINICAL TRIAL: NCT00604942
Title: Volume Sensitive Multichannel Intraluminal Impedance (vMII) for the Measurement of Oesophageal Bolus Transport and Reflux
Brief Title: vMII for Measurement of Oesophageal Bolus Transport and Reflux
Acronym: vMII
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: prototype catheter never delivered
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Dr Mark Fox, Guy's and St Thomas' NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 07/H0802/73
Record Dates: First submitted 2008-01-15; First posted 2008-01-30 (Estimated); Last update posted 2009-08-03 (Estimated); Status verified 2009-07

CONDITIONS: Achalasia; GORD
Keywords: Oesophagus; Dysphagia; Impedance; High Resolution Manometry; Peristalsis; Contractile Pressure; Coordination of contraction; Bolus transport
MeSH Terms: conditions — Esophageal Achalasia; Deglutition Disorders | interventions — Heller Myotomy; Fundoplication; Domperidone; Esomeprazole; Conservative Treatment

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Achalasia (Experimental): Long vs Short Myotomy repair of Achalasia
  Interventions: Procedure: Heller's Myotomy
- Dysphagia control (Experimental): Conservative Management
  Interventions: Drug: domperidone or esomeprazole (Conservative management)
- GORD for surgery (Experimental): Partial vs Full Fundoplication repair
  Interventions: Procedure: Nissen Fundoplication
- GORD not for surgery (Experimental): esomeprazole 40 mg vs no esomeprazole
  Interventions: Drug: Esomeprazole 40 mg

INTERVENTIONS:
Procedure: Heller's Myotomy — Long vs Short Heller's Myotomy for Achalasia
  Arms: Achalasia
Procedure: Nissen Fundoplication — Partial vs Full Fundoplication for GORD
  Arms: GORD for surgery
Drug: domperidone or esomeprazole (Conservative management) — Conservative management for dysphagia not referred for surgery. Conservative management: balloon dilatation or drugs such as domperidone 10 mg or esomeprazole 40 mg
  Arms: Dysphagia control
Drug: Esomeprazole 40 mg — Esomeprazole vs no esomeprazole for GORD not referred for surgery
  Arms: GORD not for surgery

SUMMARY:
Recent work at St. Thomas' has validated an innovative new design of a multichannel intraluminal impedance (MII) catheter that is sensitive to variation in oesophageal volume in healthy volunteers and patients. This project will establish the clinical value of volume sensitive MII (vMII) compared to conventional MII acquired simultaneously by the same catheter (ROC analysis). Studies will assess:

1. The accuracy of volume measurements and correlation between symptoms and the volume of bolus retention in patients with dysphagia.
2. The accuracy of volume measurements and correlation between symptoms and reflux volume in patients with reflux disease.

Follow up studies after appropriate treatment will assess whether symptomatic improvement is associated with a reduction in oesophageal volume retention/reflux.

The vMII technique will be applied with high resolution manometry (HRM). These investigations are complementary in that vMII assesses the success or failure of bolus transport (or occurrence of reflux) and HRM can assess:

1. the oesophageal dysfunction that results in bolus escape
2. the abnormal events at the gastro-oesophageal junction (reflux barrier) that allow reflux to occur.

with a reduction in oesophageal volume retention / reflux.

DETAILED DESCRIPTION:
Swallowing problems and gastro-oesophageal reflux disease (GORD) are common in the community with important effects on health, quality of life and NHS costs. Furthermore, these problems may explain the increasing rate of oesophageal cancer. These concerns highlight the importance of appropriate investigation and management of these symptoms.

Medications that suppress gastric acid relieve symptoms in many patients; however this does not improve oesophageal function or reduce 'non-acid' reflux from the stomach. At least 1 in 4 patients have symptoms despite treatment and further management of these individuals is challenging. Conventional multichannel intraluminal impedance (MII) studies assess swallowing function and reflux, but cannot assess volume. This is important because larger volumes of food stuck in the oesophagus and failure to clear larger amounts of irritant reflux from the stomach are more likely to cause symptoms and damage to the lining of the oesophagus.

The proposed project builds on recent work at St. Thomas' in which a new MII technique was shown to detect changes in oesophageal volume. The aim is to assess whether this volume sensitive MII (vMII) is useful in clinical practice.

Patients with swallowing problems and reflux symptoms will undergo vMII and High Resolution Manometry in unison in a combined Catheter Assembly during a test meal containing barium (known as videofluoroscopy) as it is visible on x-ray. The volume of fluid stuck in the oesophagus or refluxing from the stomach will be measured by both vMII and videofluoroscopy and the problems with motility will be assessed with HRM. The results will be compared and the link between oesophageal volume, dysmotility and symptoms will be examined. Finally the studies will be repeated after treatment (videofluoroscopy being offered only males and women over 40) to see if improvements are linked to reduced volume measurements.

In routine clinical practice, successful vMII would reduce the need for barium swallows (therefore reducing exposure to radiation) and improve the ability to link oesophageal dysfunction and reflux events with symptoms, and thus guide further management in patients that fail to respond to standard treatments.

Existing measurements of oesophageal function assess the presence or absence of acid (pH), bolus transport (HRM) or fluid (conventional MII) in the oesophagus, but are not sensitive to volume change. It is thought that this explains the failure to establish the cause of oesophageal symptoms in some patients (Sifrim Gut 06). Firstly because retention and reflux of large volumes in the oesophagus is more likely to cause symptoms. Secondly because conventional MII lacks sensitivity in patients with poor emptying of residual fluid in the oesophagus much of the time (e.g. achalasia, post-fundoplication). Volume sensitive MII (vMII) is a novel adaptation of catheter technology that is sensitive to volume changes in the oesophagus of healthy volunteers (Fox DDW 06). It is a non disposable catheter which is 3mm in diameter and is very similar to the impedance and pH manometry catheters routinely used at St Thomas' and many other hospitals and are well tolerated by patients.

Study Design and Methodology Studies will be performed in two, well-defined patient populations that represent the two cardinal presenting symptoms in oesophageal disease.

1. Patients with swallowing difficulty (dysphagia) related to achalasia
2. Patients with reflux symptoms referred for consideration of fundoplication. Individuals (age 18-65 years) referred to the oesophageal laboratory for investigation will be invited to participate. All participants will undergo complete physical and mental health questionnaires, and an assessment of predominant complaint and symptom severity.

This study will test two key issues in order to compare the clinical value of volume measurements by vMII to existing techniques in these two patient populations.

1. Stationary: The accuracy of volume measurements acquired by vMII in patients with oesophageal disease compared to videofluoroscopy (gold standard).
2. Ambulatory: The association of volume measurements with symptoms compared to conventional pH / MII measurements before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* male or female
* at least 18 years of age
* have given informed consent for the vMII and Barium videofluoroscopy
* have symptoms of reflux, dysphagia, have known achalasia or are planned for anti-reflux surgery

Exclusion Criteria:

* with medications influencing gastrointestinal function within 3 days of the study
* with those on anticoagulants
* with any hematological abnormalities
* with any evidence of infectious disease
* who are pregnant or breast-feeding or sexually active and not on contraception.
* with evidence or history of drug or alcohol abuse within the past two years
* with diabetes mellitus
* with severe physical or mental health concerns on screening which may contribute to the ability to comply with study requirements
* with active co-morbid conditions
* with oesophageal surgery or stent (dilation acceptable)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2007-11; Primary Completion 2010-10 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
Does vMII provide an accurate assessment of volume in disease? | 3 years
Does vMII assessment of volume improve the accuracy with which 'events' are associated with symp? | 3 years
Does symp improvement post treatment correlate with reduced 'volume events'?. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Mark Fox, MD, Principal Investigator — Honorary Consultant and Senior Lecturer
Locations (1):
- Oesophageal Laboratory, GSTT, London, London, United Kingdom